CLINICAL TRIAL: NCT00634647
Title: A Phase II Study of Satraplatin and Prednisone in Metastatic Androgen Independent Prostate Cancer (AIPC)
Brief Title: Satraplatin and Prednisone to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Dahut Jr., M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080074; 08-C-0074
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer; Genetic Polymorphism
Keywords: Chemotherapy; Pharmacokinetics; Gene Polymorphisms; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — satraplatin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Satraplatin (Experimental): satraplatin - 80 mg/m^2 days 1-5 of every 35 day cycle prednisone - 5 mg twice daily every 35 days
  Interventions: Drug: Satraplatin; Drug: prednisone

INTERVENTIONS:
Drug: Satraplatin — 80 mg/m^2 days 1-5 of every 35 day cycle
Drug: prednisone — 5 mg twice daily every 35 days

SUMMARY:
Background:

Satraplatin is an experimental drug that may be of benefit to patients with prostate cancer.

Prednisone is approved for treating prostate cancer.

The gene excision repair cross-complementing rodent repair deficiency complementation group 1 (ERCC1) helps repair cell damage caused by satraplatin. It is possible that patients who have a variant of this gene will not benefit from treatment with satraplatin because the drug will not be able to damage the cancer cells effectively.

Objectives:

To determine if satraplatin may help treat prostate cancer in patients with certain variants of the ERCC1 gene.

Eligibility:

Patients with advanced androgen-independent prostate cancer whose disease has not responded to hormonal therapy or at least one type of chemotherapy and whose x-rays, scans or other tests have shown their cancer to be spreading.

Design:

Participants have a blood test to determine if they have a variant of the ERCC1 gene.

Participants take satraplatin by mouth every day for 5 consecutive days out of every 35 days and prednisone by mouth every day. These 35-day treatment cycles may continue for 6 months or longer, depending on the benefits and side effects of the treatment.

During the treatment period, patients undergo the following tests and procedures:

* Blood tests on days 1 of the treatment cycle.
* Weekly blood draws for the first 3 treatment cycles.
* Imaging studies (e.g., bone scans, computed tomography (CT) scans) every two cycles to determine the response to treatment.
* Surgical or medical suppression of testosterone in patients whose cancer cells continue to grow due to exposure to the hormone....

DETAILED DESCRIPTION:
Background:

* Satraplatin is an oral, third-generation platinum analog that has recently been shown to increase prostatic specific antigen (PSA) decline rates and progression-free survival in hormone-resistant prostate cancer.
* Satraplatin acts by binding to deoxyribonucleic acid (DNA) forming intra- and interstrand cross links (DNA adducts), resulting in cell-cycle arrest in G2 phase and eventual apoptosis. One of the mechanisms that bring about resistance to platinum-based chemotherapy is removal of the platinum-DNA adducts by DNA repair pathways, called nucleotide excision repair (NER) and base excision repair (BER) pathways.
* Polymorphisms in the DNA repair genes causing impaired NER and BER capability has recently been shown in some cancers, including head and neck squamous cell carcinoma, non-small cell lung carcinoma, and ovarian carcinoma to predict better treatment outcome and response to platinum treatment.

Objectives:

* Primary objective of this single arm study is to determine if the presence of ERCC1 variant gene polymorphism which is involved with DNA damage repair may be associated with an impact on the progression-free survival of patients with metastatic prostate cancer.
* Secondary objectives of this study includes demonstration of biologic effect by the drug satraplatin in the patient and in the tumor whenever possible, by obtaining tissue biopsy and white blood cell collections, to determine correlation of biologic or clinical effects with PSA progression, evaluate correlations between genotype expression, repair pathways and clinical events, and obtain laboratory correlates which will include pharmacogenetic analysis of prostate cancer patients with genotyping using Polymerase chain reaction (PCR) followed by either restriction fragment length polymorphism or direct sequencing to genotype single nucleotide polymorphisms of ERCC1, x-ray repair cross-complementing protein 1 (XRCC1), and poly (ADP-ribose) polymerase 1 (PARP1).

Eligibility:

* Patients with metastatic androgen-independent prostate cancer.
* Had docetaxel-based chemotherapy, but no more than 1 previous cytotoxic chemotherapy line.
* Good organ function.

Design:

* Phase II trial with single stage design and a planned accrual of 66 patients.
* Progression-free survival will be determined using a Fisher's exact test.
* Will treat all enrolled patients with oral satraplatin 80 mg/m^2 dose on days 1-5 of every 35-days cycle plus Prednisone 5 mg twice daily every 35 days.
* Genotyping will be performed after the first 20 patients to determine if the proportion for wild-type ERCC1 and variants follow a 20:80 split.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Patients must have histopathological confirmation of prostate cancer by the Laboratory of Pathology of the National Cancer Institute (NCI) or Pathology Department of the National Naval Medical Center or Walter Reed Army Medical Center prior to entering this study. Patients whose pathology specimens are not available may be enrolled in the trial if the patient has a clinical course consistent with prostate cancer and available documentation from an outside pathology laboratory of the diagnosis. In cases where original tissue blocks or archival biopsy material is available, all efforts should be made to have the material forwarded to the research team for use in correlative studies.

B. Patients must have metastatic progressive androgen-independent prostate cancer. There must be radiographic evidence of disease (by computed tomography (CT) scan or bone scan) after primary treatment that has continued to progress despite hormonal agents. Progression requires that a measurable lesion is expanding, new lesions have appeared, and/or that prostatic specific antigen (PSA) is continuing to rise on successive measurements. Patients must have progressive disease after receiving 1 prior docetaxel-based cytotoxic chemotherapy. Patients on flutamide for the prior 6 months must have disease progression at least 4 weeks after withdrawal. Patients on bicalutamide or nilutamide must have progression at least 6 weeks after withdrawal.

C. Patients may only have received 1 prior cytotoxic chemotherapy. For the purpose of this study, multiple courses of a taxane-based regimen may count as a single regimen. Multiple courses of a non-taxane agent or a combination chemotherapy regimen, administered in a similar fashion may count as a single regimen.

D. Patients must have a life expectancy of more than 3 months.

E. Patients must have a performance status of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) criteria.

F. Patients must have adequate organ function as defined below:

Leukocytes greater than or equal to 3,000/microl.

Absolute Neutrophil Count greater than or equal to 1,500/microl.

Platelets greater than or equal to 100,000/microl.

Total bilirubin less than or equal to 1.5 times institutional upper limits of normal (Except patients with Gilbert's disease who may proceed despite elevated total bilirubin).

Aspartate aminotransferase (AST)serum glutamic oxaloacetic transaminase(SGOT) and alanine aminotransferase (ALT)serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times institutional upper limit of normal

Creatinine less than or equal to 1.5 times institutional upper limits of normal.

OR

Creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

G. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be <= grade 1 or returned to baseline.

H. Hormonal profile: all patients who have not undergone bilateral surgical castration must continue suppression of testosterone production by appropriate usage of gonadotropin releasing hormone (GnRH) agonists.

I. Patients must not have any ongoing malignancies requiring active therapy.

J. Patients must be able to understand and sign an informed consent form.

K. Concurrent use of bisphosphonates will be allowed if patients have previously been on it; if patients are not on bisphosphonates at the time of study enrollment, bisphosphonates may be started at cycle 2.

L. Patients who require hematopoietic growth factor support (e.g. epogen, darbepoetin), but not myeloid growth factors (except after cycle 1 day 1 if clinically indicated), non-steroidal anti-inflammatory drug (NSAIDs), and other maintenance medications prior to study entry will be allowed to continue their supportive therapies.

M. Results from embryo-fetal development indicated that satraplatin should be considered a teratogen in women of childbearing potential and hazardous in respect to spermatogenesis for men. For this reason, men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.

N. Patients must be able to swallow capsules.

O. Patients on chronic stable steroids (equivalent to no more than 10 mg of prednisone daily dose) used for non-cancer treatment may be allowed on study.

EXCLUSION CRITERIA:

A. Patients who have had prior treatment with satraplatin or other platinum containing compounds will be excluded.

B. Patients may not be receiving any other investigational agents.

C. Patients with known active brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

D. History of allergic reactions attributed to compounds of similar chemical or biologic composition to satraplatin or prednisone.

E. Uncontrolled intercurrent illness including, but not limited to ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit patient compliance with study requirements.

F. Prior radiation therapy to greater than 30 percent of the bone marrow, or who have received strontium-89, rhenium-186, or rhenium-188 will be excluded from this trial. Patients who have received prior radiotherapy must have recovered from acute toxicity due to radiation. Patients who have received samarium-153 are eligible for the study because samarium has a significantly reduced half-life compared to aforementioned isotopes.

G. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, human immunodeficiency virus (HIV)-positive patients are excluded from the study.

H. Patients with a history of major gastrointestinal surgery or pathology likely to influence absorption of oral medications, like bypass surgeries, Whipple's procedure, or any surgery that would impair reliable absorption of oral drugs.

I. Patients with a disease where corticosteroids are contraindicated, e.g. active gastric or duodenal ulcer, or poorly controlled insulin dependent diabetes. Patients with well-controlled insulin-dependent diabetes mellitus may be considered, providing they understand their glucose levels will increase, and their insulin dose will require adjusting.

J. Because no dosing or adverse event data are currently available on the use of satraplatin in patients less than 18 years of age, children are excluded from this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02-19 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2012-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Associates in Oncology and Hematology, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moul JW. Prostate specific antigen only progression of prostate cancer. J Urol. 2000 Jun;163(6):1632-42. PMID 10799151
- [Background] Zelefsky MJ, Ben-Porat L, Scher HI, Chan HM, Fearn PA, Fuks ZY, Leibel SA, Venkatraman ES. Outcome predictors for the increasing PSA state after definitive external-beam radiotherapy for prostate cancer. J Clin Oncol. 2005 Feb 1;23(4):826-31. doi: 10.1200/JCO.2005.02.111. PMID 15681527
- [Background] Catalona WJ, Smith DS. Cancer recurrence and survival rates after anatomic radical retropubic prostatectomy for prostate cancer: intermediate-term results. J Urol. 1998 Dec;160(6 Pt 2):2428-34. doi: 10.1097/00005392-199812020-00012. PMID 9817397
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0074.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Satraplatin
Started | 24
Completed | 17
Not Completed | 7
Not completed — death on study | 3
Not completed — refused further treatment | 3
Not completed — declined to participate before treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Satraplatin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.83 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival.
Description: Time between the start of therapy and progression. Progression is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Progressive Disease is at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 15 months
Population: 24 pts were enrolled but only 21/24 were assessed for OS. One pt died on treatment and (e.g.3 pts were non-evaluable for analysis of response).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Satraplatin
Number analyzed (Participants) | 20
Months | 6.0 [2.3 to 9.3]

2. Secondary Outcome: Number of Participants With Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 57 months.
Population: The time frame for adverse events includes one year follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Satraplatin
Number analyzed (Participants) | 23
Participants | 23

3. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival is the time between the first day of treatment to the day of death.
Time Frame: time between the first day of treatment to the day of death, approximately 15.7 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Satraplatin
Number analyzed (Participants) | 21
Months | 16.0 [6.5 to NA] — The upper limit of the confidence interval was not reached because patients were on-study at the time data was analyzed.

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 57 months.
Description: The time frame for adverse events includes one year follow-up data.
Arm/Group | Satraplatin
All-Cause Mortality (participants affected / at risk) | 11/23
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Satraplatin (N=23)
Hemoglobin (Blood and lymphatic system disorders) | 1 (2)
Infection, Other (septic shock) (Infections and infestations) | 1 (2) — patient died from septic shock
Pain (General disorders) | 1 (1) — pain
Platelets (Blood and lymphatic system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Death (General disorders) | 10 (10) — 2 patients died from progressive disease and 8 died in follow-up from progressive disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Satraplatin (N=23)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (6)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 8 (9)
Alkaline phosphatase (Metabolism and nutrition disorders) | 8 (10)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 6 (6)
Bicarbonate, serum low (Metabolism and nutrition disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (6)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6)
Creatinine (Metabolism and nutrition disorders) | 3 (3)
Dental: periodontal disease (Gastrointestinal disorders) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 1 (1)
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 2 (2) — left ear "blk lesion" papular flat; rashes
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (9)
Fever (General disorders) | 1 (2) — (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Flu-like syndrome (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal-Other (pain intermittent diarrhea) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 15 (25)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder tract NOS (Infections and infestations) | 1 (3)
Insomnia (General disorders) | 3 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 15 (38)
Lymphopenia (Blood and lymphatic system disorders) | 14 (25)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 4 (4)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 4 (4)
Mucositis/stomatitis (clinical exam)::oral cavity (Gastrointestinal disorders) | 1 (1)
Musculoskeletal/soft tissue-Other, muscle cramping (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (11)
Neuropathy:sensory (Nervous system disorders) | 3 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 12 (21)
Ocular/Visual-Other, visual field deficit (blind spot) (Eye disorders) | 1 (1)
Pain -Other,intermittent LE pain (General disorders) | 1 (1)
Pain-abdomen NOS (Gastrointestinal disorders) | 2 (3)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain::Pelvis (Reproductive system and breast disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (7)
Platelets (Blood and lymphatic system disorders) | 18 (51)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 (8)
Renal failure (Renal and urinary disorders) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2011-05-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT00634647/Prot_ICF_000.pdf